CLINICAL TRIAL: NCT05697601
Title: Associated Factors of Ovarian Cancer and Endometrial Cancer in Indonesia. A Study for Developing Artificial-Intelligence-Based Screening Tools
Brief Title: Predictors of Ovarian Cancer and Endometrial Cancer for Artificial-Intelligence-Based Screening Tools
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hasanuddin University (Other)
Collaborators: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Bumi Herman, Assistant Lecturer, Hasanuddin University
Other Study IDs: 0901231327
Record Dates: First submitted 2023-01-14; First posted 2023-01-26 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Ovarian Cancer; Endometrial Cancer; Endometrial Hyperplasia
Keywords: Ovarian Cancer; Endometrial Cancer; Endometrial Hyperplasia; Artificial Intelligence; Point of Care Testing; Staging; Gynecological Screening; Pathology
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Endometrial Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Suspect of Ovarian Cancer: The participant with high suspicion of ovarian cancer and undergo gynaecology and pathology assessment
  Interventions: Diagnostic Test: Artificial-Intelligence Based Screening Tools; Diagnostic Test: Pathology analysis
- Suspect of Endometrial Cancer: The participant with high suspicion of Endometrial cancer (and or endometrial hyperplasia) and undergo gynaecology and pathology assessment
  Interventions: Diagnostic Test: Artificial-Intelligence Based Screening Tools; Diagnostic Test: Pathology analysis
- Normal Cohort: The participant with lower suspicion of both types of cancer and undergo gynaecology and pathology assessment
  Interventions: Diagnostic Test: Artificial-Intelligence Based Screening Tools; Diagnostic Test: Pathology analysis

INTERVENTIONS:
Diagnostic Test: Artificial-Intelligence Based Screening Tools — Artificial-Intelligence Based Screening Tools build on machine learning models
Diagnostic Test: Pathology analysis — Pathology assessment of cells and tissues from respective organs

SUMMARY:
The goal of this observational study is to explore the possible associated factors of ovarian cancer and endometrial cancer in Indonesia and develop screening tools that could predict the risk of both types of cancer

The specific objectives of the study are

1. Elaborating the situation of ovarian and endometrial cancer in Indonesia
2. Exploring the possible clinical, demography and laboratory predictors of these diseases
3. Develop artificial-intelligence-based screening tools for both type of cancer based on possible predictors

This study will utilize the patient registry diagnosed with ovarian and endometrial cancer. We assumed that several demography, clinical, and laboratory predictors might possess good screening performance with higher sensitivity and specificity (>80%).

DETAILED DESCRIPTION:
Methodology :

This study will involve two different stages

1. The first stage will conduct a cohort study to identify the possible predictors of each type of cancer
2. The second stage will cover the development of point-of-care testing based on an artificial intelligence model to predict cancer occurrence and prospective testing of the new participants using a diagnostic study method. The tools will predict the current histopathology result and possible future histopathology within one year.

Participants and source of data In the study centre, women with or without gynaecology-associated symptoms underwent gynaecological and pathology assessments to rule out ovarian and endometrial cancer in our study centre were involved. Data is stored digitally and extraction will be done accordingly

Variables and outcome measurement

1. Demographic data and health data this information is obtained from the initial assessment of the patients including age, body mass index, chronic diseases, gynaecological and obstetric profile, menstrual pattern, and contraception
2. Clinical and laboratory data this include, a complete blood count, selected cancer-associated biomarker (for example Cancer Antigen 125 (Ca-125)), involvement of lymph node, histopathology of pertinent tissues, and signs of metastases through clinical or radiological data
3. Outcome final histopathology type and classification assessed by at least two pathologists to determine the type of cancer. The guidelines of classification follow the World Health Organization's classification

Development of Artificial-Intelligence-based screening tools

1. The researcher will develop

   - an information-based model where the user will provide a response to each predictor

   - an image-based model where the user will provide a captured image for prediction

   - a mixed-based model where the user can combine captured images and information for each predictor
2. proposed model

   - scoring-based derived from the coefficient of regression

   - decision tree

   - random forest

   - artificial neural network
   * convolutional neural network
3. Selection of model

<!-- -->

1. Screening performance on split data (or using cross-validation technique)
2. evaluation of log-loss or likelihood

   Timeline

   1. For the first stage of the study, there will be a time-varying assessment for each participant, however, at least participants undergo an Assessment of all factors and outcomes at baseline. Repeated evaluation as suggested by the physician will be done within one year after the baseline assessment.

   2. The second study will apply prospective screening. The artificial intelligence-based screening tool will be used concurrently with the gold standard of diagnosis.

   Possible Bias procedural bias particularly in reliability outcome interpretation is handled by involving multiple pathologists. The pathologist and the screener will perform the screening independently to reduce the tendency of prior results provided by the newly-developed screening tools.

   Sample size
   1. The first stage of the research assumes that

a. The prevalence of both cancer among all cancers in women accounted for 5% b. Type I error set at 5% c. absolute error of the prevalence 1% using the one-sample proportion formula, the estimated sample size is 1825 participants.

2. Following the diagnostic study, we state that the new screening tools model will show non-inferiority performance to histopathology as gold-standard, assuming that

a. the expected difference in sensitivity value is 5% assuming that the new screening tools will possess 85% sensitivity and the sensitivity of histopathology is 90% b. cross-over testing will be done, creating an equal allocation of screening intervention c. Type 1 error of the study set at 5% d. Power of the study set at 80% the total sample size for the prospective screening tool will be 1080 participants

Data Quantification and discretization several clinical information will be classified according to the established guideline for example body mass index.

Proposed Statistical Analysis

1. Descriptive statistic and bivariate analysis
2. A cox-regression will be conducted following the baseline-to-event timeline
3. Subgroup analysis will be done, particularly in certain demographic and comorbidity.

as for the second stage, the analysis will identify the

1. sensitivity
2. specificity
3. accuracy
4. precision
5. The number Needed to Treat selected models will be deployed into an application.

ELIGIBILITY:
Inclusion Criteria:

* Women with gynaecological symptoms but not limited to

  1. Irregular menstruation
  2. Heavy bleeding during menstruation
  3. pelvic pain
  4. vaginal discharge
  5. sudden weight loss
  6. pain during sexual intercourse
* Women who underwent routine gynaecological examination

Exclusion Criteria:

* unable to undergo serial gynaecological follow-up

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — as the disease affects natural-born women, therefore, only women will be included
Study Population: As this study is utilizing a patient registry, we will involve all eligible participants who undergo gynaecological and pathology assessment for ovarian and endometrial cancer in study centres, based on suggestive signs and symptoms
Sampling Method: Non-Probability Sample
Enrollment: 2905 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of People developing ovarian cancer | from baseline to twelve month after entering cohort
  Number of people developing ovarian cancer diagnosed with gynaecology and pathology assessment
Number of People developing endometrial cancer | from baseline to twelve month after entering cohort
  Number of people developing endometrial cancer diagnosed with gynaecology and pathology assessment

SECONDARY OUTCOMES:
Screening Performance of Artificial-Intelligence-based Screening tools | from baseline assessment up to one year
  The sensitivity, specificity, accuracy, precision of selected Artificial-Intelligence-based model to predict the ovarian and/or endometrial cancer

CONTACTS AND LOCATIONS:
Overall Officials: Rina Masadah, Ph.D, Study Chair — Hasanuddin University; Bumi Herman, Ph.D, Principal Investigator — Chulalongkorn University
Locations (1):
- Hasanuddin University Hospital, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No
The individual participant data will be shared after de-identification and the purpose of the data utilization is verified by the investigators

REFERENCES:
- [Background] Atallah GA, Abd Aziz NH, Teik CK, Shafiee MN, Kampan NC. New Predictive Biomarkers for Ovarian Cancer. Diagnostics (Basel). 2021 Mar 7;11(3):465. doi: 10.3390/diagnostics11030465. PMID 33800113
- [Background] Elias KM, Guo J, Bast RC Jr. Early Detection of Ovarian Cancer. Hematol Oncol Clin North Am. 2018 Dec;32(6):903-914. doi: 10.1016/j.hoc.2018.07.003. Epub 2018 Sep 28. PMID 30390764
- [Background] Tanha K, Mottaghi A, Nojomi M, Moradi M, Rajabzadeh R, Lotfi S, Janani L. Investigation on factors associated with ovarian cancer: an umbrella review of systematic review and meta-analyses. J Ovarian Res. 2021 Nov 11;14(1):153. doi: 10.1186/s13048-021-00911-z. PMID 34758846
- [Background] Zhao J, Hu Y, Zhao Y, Chen D, Fang T, Ding M. Risk factors of endometrial cancer in patients with endometrial hyperplasia: implication for clinical treatments. BMC Womens Health. 2021 Aug 25;21(1):312. doi: 10.1186/s12905-021-01452-9. PMID 34433451
- [Background] Felix AS, Weissfeld JL, Stone RA, Bowser R, Chivukula M, Edwards RP, Linkov F. Factors associated with Type I and Type II endometrial cancer. Cancer Causes Control. 2010 Nov;21(11):1851-6. doi: 10.1007/s10552-010-9612-8. Epub 2010 Jul 14. PMID 20628804
- [Background] Herman B, Sirichokchatchawan W, Pongpanich S, Nantasenamat C. Development and performance of CUHAS-ROBUST application for pulmonary rifampicin-resistance tuberculosis screening in Indonesia. PLoS One. 2021 Mar 25;16(3):e0249243. doi: 10.1371/journal.pone.0249243. eCollection 2021. PMID 33765092